CLINICAL TRIAL: NCT01392014
Title: Effectiveness of Dihydroartemisinin-piperaquine With or Without Primaquine on Gametocytes Plasmodium Falciparum in Mesoendemic Area of Indonesia
Brief Title: Dihydroartemisinin-piperaquine and Primaquine for Uncomplicated Plasmodium Falciparum Cases
Acronym: DHP+PQ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Dr. Inge Sutanto, Parasitologi Fakultas Kedokteran, University of Indonesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 45114; 45114 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2011-06-24; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2008-08

CONDITIONS: Malaria
Keywords: malaria; DHP; PQ; gametocytes
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dihydroartemisinin-piperaquine (Active Comparator)
  Interventions: Drug: dihydroartemisinin-piperaquine
- Dihydroartemisininpiperaquine primaquine (Active Comparator)
  Interventions: Drug: dihydroartemisinin-piperaquine + primaquine

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine — This study used fixed-dose tablets of 40 mg dihydroartemisinin and 320 mg piperaquine for each tablet (D-ARTEPP®, Guilin Pharmaceutical Co., Ltd, China. The regimen is based on weight for 3 days (D0, D1 and D2) with maximal dose of 1 x 3 tablets for patients weighing ≥ 41 kg; 1 x 2 tablets for patients weighing 31 - 40 kg, 1 x 1.5 tablets for patients weighing 18 - 30 kg, and 1 X 1 tablet for patients with body weight of 11 - 17 kg.
  Other Names: DHP
  Arms: dihydroartemisinin-piperaquine
Drug: dihydroartemisinin-piperaquine + primaquine — For DHP, treatment was as for Arm dihydroartemisinin piperaquine. A single dose PQ of 0.75 mg/kg BW was provided on Day-3 using 15 mg base PQ tablets (local product by PT Pharos Indonesia, batch no 15306002, produced on 30/05/2008 and expiring on May 2012). The maximal dose was 3 tablets for subjects weighing ≥ 60 kg. The dose range for subjects weighing 10 - 13 kg was 0.5 tablet; 14 - 18 kg was 0.75 tablet; 19 - 23 kg was 1 tablet, 24 -30 kg was 1.5 tablet; 31 - 40 kg was 2 tablets; 41- 49 kg was 2.25 tablet; 50 - 59 kg was 2.5 tablet and ≥ 60 kg was 3 tablets.
  Other Names: DHP, PQ
  Arms: Dihydroartemisininpiperaquine primaquine

SUMMARY:
Artemisinin-based combination therapy (ACT) has been known to be controversial for stopping malaria transmission.The addition of primaquine (PQ) - the only drug commercially available that kills mature transmission stage - to such treatments might be necessary to eliminate this stage. A study is conducted to evaluate the efficacy of dihydroartemisinin-piperaquine (DHP) regimens with or without PQ on the sexual and asexual stages of P. falciparum in Sumatra, Indonesia.

DETAILED DESCRIPTION:
The study was conducted in Hanura Primary Health Center, Padang Cermin district, Lampung province (105°45'-103°48'E and 3°45'-6°45'S) located at the southern end of Sumatra island.

The study subjects received either 3 day doses of dihydroartemisinin-piperaquine with or without 1 day of primaquine according to their body weight.

Patients with fever or history of fever within the past 24 hours were screened by microscopic examination of Giemsa-stained thick blood films to detect P. falciparum infection.

All subjects were allocated by open-label randomization to receive DHP alone (on Day 0 to Day 2) or DHP plus a single dose of PQ (Day 3). The procedures of drug administration in the study were as follows:

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 4 years old
* parasite count ≥ 1,000 asexual parasites/µL
* normal glucose-6-phosphate dehydrogenase enzyme level based on qualitative test (Trinity Biotech® no 203, USA)
* hemoglobin level ≥ 8 gr/dL as measured by Hemoque® apparatus;
* have the ability to return for 42-day-follow up and
* willingness to sign the informed-consent form.

Exclusion Criteria:

* are infected with other r plasmodium species
* have only gametocytes of P. falciparum;
* are pregnant - measured by positive result on HCG urine test and/or breastfeeding women
* present signs of pitting edema on both legs as a sign of malnutrition
* have complicated or severe malaria, other chronic diseases or history of drug allergies.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Development of sexual stages of P.falciparum | 42 days post treatment
  Finger prick blood samples are collected for malaria blood smear. Thick and thin blood smears were stained with 3% Giemsa solution for 40 minutes and were read under binocular microscope with 1,000X magnification.

SECONDARY OUTCOMES:
Clearance of asexual stages P.falciparum | 42 days post treatment
  Finger prick blood samples are collected for malaria blood smear. Thick and thin blood smears were stained with 3% Giemsa solution for 40 minutes and were read under binocular microscope with 1,000X magnification.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Sutanto, MD, Principal Investigator — Univesity of Indonesia
Locations (1):
- Hanura Primary Health Center, Lampung, Sumatra, Indonesia

REFERENCES:
- [Derived] Sutanto I, Suprijanto S, Kosasih A, Dahlan MS, Syafruddin D, Kusriastuti R, Hawley WA, Lobo NF, Ter Kuile FO. The effect of primaquine on gametocyte development and clearance in the treatment of uncomplicated falciparum malaria with dihydroartemisinin-piperaquine in South sumatra, Western indonesia: an open-label, randomized, controlled trial. Clin Infect Dis. 2013 Mar;56(5):685-93. doi: 10.1093/cid/cis959. Epub 2012 Nov 21. PMID 23175563